CLINICAL TRIAL: NCT06670066
Title: Rigorous Evaluation of Let's Talk Birth Control Among Adolescents Attending Community Health Centers
Brief Title: Rigorous Evaluation of Let's Talk Birth Control
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Child Trends (Other)
Collaborators: University of California, San Francisco (Other); Power to Decide (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TP22023001568; TP22023001568 (Other Grant/Funding Number: Office of Population Affairs)
Record Dates: First submitted 2024-10-28; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Sexual Behavior; Adolescent Behavior
MeSH Terms: conditions — Sexual Behavior; Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: This research project will use a cluster-level randomized control trial design in which a participating health center is randomized to either the experimental condition (Let's Talk Birth Control) or the control condition (standard health services). All participants enrolled at health centers randomized to the experimental condition should receive the Let's Talk Birth Control intervention while all participants enrolled at health centers randomized to the control condition should receive health services as usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adolescents receiving Let's Talk Birth Control (Experimental): Participants in the Let's Talk Birth Control condition receive access to the CDA materials, contraceptive counseling with trained healthcare providers, and asynchronous access to the Bedsider ME web platform.
  Interventions: Behavioral: Let's Talk Birth Control
- Adolescents receiving standard reproductive and sexual health care services (No Intervention): Participants in the control condition receive standard health care services from their medical provider. Health centers in the control condition will not be using an adolescent-focused sexual and reproductive health CDA or contraceptive counseling initiative.

INTERVENTIONS:
Behavioral: Let's Talk Birth Control — Let's Talk is an innovative, multi-level intervention addressing adolescents and providers that includes both in-person and online components and is feasible to implement in clinical settings. The three core components are: (1) a printed contraceptive decision aid (CDA) with a QR code linking to the Method Explorer (ME) page on Power to Decide's online birth control website, Bedsider; (2) the Bedsider ME, with information on the full range of contraceptive methods and a personalized method comparison feature; and (3) an online training for providers on Patient-centered Contraceptive Counseling (PCCC), including use of the CDA to support shared decision-making with adolescents.
  Arms: Adolescents receiving Let's Talk Birth Control

SUMMARY:
The goal of this cluster-level randomized controlled trial is to evaluate the impacts of Let's Talk Birth Control, a clinical decision support intervention for adolescents that consists of a printed contraceptive decision aid (CDA), contraceptive counseling, and a QR code to the Bedsider.org Method Explorer (ME). The goal of Let's Talk Birth Control is to reduce rates of sex without a contraceptive method among adolescent patients, increase use of preferred contraceptive method, as well as to increase self-efficacy to discuss, obtain, and correctly use contraceptive methods

The primary research questions are:

* Does receiving care from a health center participating in Let's Talk Birth Control reduce rates of sex without a contraceptive method among adolescent patients compared to those visiting a standard of care control health center?
* Does receiving care from a health center participating in Let's Talk Birth Control increase use of preferred contraceptive method among adolescent patients compared to those visiting a standard of care control health center?

The evaluation will focus on the impacts of receiving the Let's Talk Birth Control intervention, as compared to receiving standard health care services.

As part of this study:

* All participants will be asked to complete baseline, 1-week post-intervention, and 9-month follow-up surveys.
* Participants at health centers randomized to receive the Let's Talk intervention, will be asked to:
* Review the Let's Talk CDA independently prior to meeting with their healthcare provider
* Participate in an observation focused on the provider's use of the CDA for contraceptive counseling during the healthcare visit (select participants only)
* Participate in a focus group discussing their perceptions of the Let's Talk Birth Control intervention (select participants only)

Staff at health centers randomized to receive the Let's Talk intervention will be asked to:

* Complete a 45-60 minute online asynchronous training covering patient-centered contraceptive counseling (PCCC) for adolescents and using the CDA
* Use the Let's Talk CDA to facilitate patient-centered contraceptive counseling with patients that have enrolled in the study

ELIGIBILITY:
Inclusion Criteria:

Health Centers:

* Serve 400+ patients assigned female at birth (AFAB) aged 15-24 receiving sexual and reproductive health (SRH) services or general wellness exams annually. Although the project team may enroll rural health centers with smaller populations
* Have not implemented an adolescent SRH patient-centered training recently
* Do not utilize a contraceptive decision aid (CDA) designed for adolescent patients

Participants:

* Assigned female at birth
* Seeking sexual and reproductive services or general wellness exams at an enrolled community health center
* Have had penile-vaginal sex in the past year or are interested in discussing birth control with their provider
* Agree to be in study

Exclusion Criteria:

Health Centers

* Does not serve at least 400 AFAB aged 15-24 receiving SRH services or general wellness exams annually
* Has recently implemented an adolescent SRH training
* Currently using a CDA designed for adolescent patients

Participants:

* Does not agree to be in study
* Is pregnant or is trying to become pregnant
* Does not have access to a phone to receive text messages
* Does not speak English or Spanish

Ages: 15 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1500 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Rates of sex without a contraceptive method | 9 months post-intervention
  Penile-vaginal sex without any contraception (including condom) in the past 3 months (yes/no).
  Yes if had sex in the past 3 months and did not use a contraceptive method "all the time". No if did not have sex or used a contraceptive method "all the time".
Use of preferred contraceptive method | 9 months post-intervention
  Currently using preferred birth control method (yes/no). Respondents are coded as No if they report there is a method of birth control that they would like to be using right now but are not currently using. Otherwise, they are coded as Yes.

SECONDARY OUTCOMES:
Self-efficacy to discuss contraception with a provider | 1 week post-intervention
  Confident they can talk about birth control with their doctor or health care provider (yes/no, "Strongly agree" vs other responses).
Self-efficacy to make informed decisions about contraception | 1 week post-intervention
  Strongly agree that they 1) feel sure about the best birth control option for their needs and 2) have received enough support and advice to make a choice about birth control methods (yes/no, "Strongly agree" to both items vs other responses)
Intentions to use contraception | 1 week post-intervention
  Intends to use contraception if chooses to have penile-vaginal sex in the next 3 months (yes/no, "Yes, definitely" vs other responses)
Self-efficacy to use contraception | 1 week post-intervention
  4-item Likert scale capturing 1) confidence in starting a new method of birth control if they want, 2) using birth control correctly, 3) knowing the steps needed to continue a birth control method, and 4) avoiding unintended pregnancy (1-5 scale)
Knowledge of contraceptive methods | 1 week after post-intervention
  Knowledge of contraceptive methods (% correct out of 6 items)
Attitudes about contraception | 1 week post-intervention
  6-item Contraceptive Concerns and Beliefs Scale
  Citation: Rocca, C.H., Muñoz, I., Rao, L. et al. Measuring a Critical Component of Contraceptive Decision Making: The Contraceptive Concerns and Beliefs Scale. Matern Child Health J 28, 847-857 (2024).

IPD SHARING:
Plan to Share IPD: No